CLINICAL TRIAL: NCT03843060
Title: A Phase 1 Single Center Open-label, Non-randomized, Fixed Sequence Study in Healthy Volunteers to Assess the Pharmacokinetics (PK) of AZD9977 When Administered Alone and With Itraconazole
Brief Title: A Phase 1 Study to Assess the Pharmacokinetics of AZD9977 Administered Alone and in Combination With Itraconazole in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D6401C00003
Record Dates: First submitted 2019-02-14; First posted 2019-02-15 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: Congestive heart failure; Healthy volunteers; Itraconazole; Drug-drug interaction; Pharmacokinetics; Open-label non-randomized
MeSH Terms: conditions — Heart Failure | interventions — AZD9977; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single AZD9977 (Experimental): During this treatment period, healthy participants will be administered with a single AZD9977 (Dose 1) dose, in the fed state, on Day 1 followed by at least 3 days washout period.
  Interventions: Drug: AZD9977
- Itraconazole + AZD9977 (Experimental): During this treatment period, healthy participants will be administered with Itraconazole (Dose 2) from Day 4 to Day 8 plus will be administrated with AZD9977 (Dose 1, fed state) as a single dose on Day 7. Dose of itraconazole will be taken at -1 hour (1 hour prior to AZD9977 dosing) when co-administered with AZD9977.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: AZD9977 — Participants will receive single AZD9977 (Dose 1) capsule orally once daily in fed state, on Day 1 followed by at least 3 days washout period.
  Arms: Single AZD9977
Drug: Itraconazole — Participants will receive Itraconazole daily (Dose 2) capsule orally once daily from Day 4 to Day 8 plus will be administered AZD9977 (Dose 1, fed state) as a single dose on Day 7. Dose of itraconazole has to be taken at -1 hour (1 hour prior to AZD9977 dosing) when co-administered with AZD9977.
  Other Names: Sporanox
  Arms: Itraconazole + AZD9977

SUMMARY:
This is an open-label, non-randomized, fixed sequence study conducted at a single study center with primary aim to assess the pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, fixed sequence study conducted at a single study center with primary aim to assess the pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole. Two types of treatments (treatment period 1 and treatment period 2) will be administered in a fixed order separated by a washout period of 3 days or more. Treatment period 1 will be single dose of AZD9977 (Dose 1) administration, in the fed state, on Day 1 followed by at least 3 days washout period. For treatment period 2, Itraconazole will be administered daily (Dose 2) from Day 4 to Day 8 plus AZD9977 (Dose 1, fed state) will be administered as a single dose on Day 7. Dose of itraconazole has to be taken at -1 hour (1 hour prior to AZD9977 dosing) when co-administered with AZD9977.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and female participants of non-childbearing potential aged 18 - 55 years with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:

   1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone (FSH) levels ≥40 mlU/ml.
   2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study..
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.

Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the PI including serum potassium > 5.0 mmol/L, serum hsTnI > 25.6 pg/mL, and NT-pro-BNP > 124 pg/mL.

5. Any clinically significant abnormal findings in vital signs as specified below and as judged by the PI at screening and on admission including:

1. Systolic blood pressure (SBP) < 90 mmHg or > 140 mmHg.
2. Diastolic blood pressure (DBP) < 50 mmHg or > 90 mmHg.
3. HR < 45 or > 90 beats per minute (bpm). 6. Any clinically significant abnormalities on 12-lead ECG, as judged by the PI.

   7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

   8. Known or suspected history of drug abuse in the last 12 months as judged by the Investigator.

   9. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.

   10. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.

   11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977.

   12. Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 3 months prior to screening.

   13. Positive screen for drugs of abuse, cotinine or alcohol at screening or on each admission to the study center.

   14. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.

   15. Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life.

   16. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol in the last 12 months as judged by the PI.

   17. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.

   18. Participants who have previously received AZD9977. 19. Judgment by the PI that the participant should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

   20. Vulnerable participants , e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

   21. Participants with any special dietary restrictions such as participants that are lactose intolerant or are vegetarians/vegans.

   22. Drugs affecting CYP3A4 (itraconazole) should be refrained from use for 3 weeks prior to study commencement and thereafter until study completion.

   23. The following exclusion criterion is driven by contraindications from the proposed concomitant CYP3A4 (itraconazole) inhibitor medications: Itraconazole (Sporanox) capsules are contra-indicated in patients with known hypersensitivity to itraconazole or to any of the excipients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUC) for AZD9977 | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast) for AZD9977 | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole
Maximum observed plasma concentration (Cmax) for AZD9977 | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole

SECONDARY OUTCOMES:
Time to reach Maximum Observed Plasma Concentration (tMax) | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole
Mean residence time of the unchanged drug in the systemic circulation from time zero to infinity (MRT) | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole.
Terminal elimination rate constant (λz) | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole
Apparent total body clearance of drug from plasmsa after extravascular administration (CL/F) | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | Day 1 to 3: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose. Day 4 to 9: pre-dose on Day 7 and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 8, 12, 16, 24, 36 and 48 hours post-dose
  To access pharmacokinetics (PK) of AZD9977 in healthy volunteers when administered alone and in combination with multiple doses of itraconazole
Number of participants with adverse events (AEs) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess AEs as variable of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal blood pressure (both systolic and diastolic blood pressure) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To measure BP as variable of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole. BP will be collected after the participants has rested in the supine position for at least 5 minutes.
Number of participants with abnormal pulse rate | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To measure pulse rate as variable of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole. Pulse rate will be collected after the participants has rested in the supine position for at least 5 minutes.
Number of participants with abnormal 12-lead Electrocardiograms (ECG) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To examine the safety and tolerability of AZD9977 in combination with itraconazole. 12-lead safety ECG will be obtained after the participant rested in the supine position for at least 10 minutes using the sites own ECG machines. The Principal Investigator (PI) will judge the overall interpretation as normal or abnormal and this evaluation will be reported in ClinBase. If abnormal, it will be further documented as to whether or not the abnormality is clinically significant by the PI.
Number of participants with abnormal physical examination findings | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess any clinically significant abnormal physical examination findings as a variable of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole. The complete physical examinations will include an assessment of the general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems. The brief physical examinations will include an assessment of the general appearance, skin, abdomen, cardiovascular system and respiratory.
Number of participants with abnormal laboratory assessments: Hematology- White blood cell (WBC) count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the white blood cell count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of participnats with abnormal laboratory assessments: Hematology- Red blood cell (RBC) count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the red blood cell count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of paticipants with abnormal laboratory assessments: Hematology - Hemoglobin (Hb) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the Hb as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of participants with abnormal laboratory assessments: Hematology - Hematocrit (HCT) and Reticulocyte absolute count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the HCT and reticulocyte absolute count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Hematology - Mean corpuscular hemoglobin (MCH) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the MCH as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Hematology - Mean corpuscular volume (MCV) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the MCV as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Hematology - Mean corpuscular hemoglobin concentration (MCHC) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the MCHC as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Hematology- Neutrophils absolute count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the neutrophils absolute count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of participants with abnotmal laboratory assessments: Hematology- Lymphocytes absolute count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the Lymphocytes absolute count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of participants with abnormal laboratory assessments: Hematology- Monocytes absolute count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the Monocytes absolute count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of participants with abnormal laboratory assessments: Hematology- Eosinophils absolute count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the Eosinophils absolute count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of participants with abnormal laboratory assessments: Hematology- Basophils absolute count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the Basophils absolute count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of participants with abnormal laboratory assessments: Hematology- Platelets count | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the Platelets count as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - Calcium, potassium, phosphate and sodium | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the serum calcium, potassium, phosphate and sodium level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - Liver enzymes | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the serum Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Aspartate aminotransferase (AST) and Gamma glutamyl transpeptidase (GGT) level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - Albumin | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the albumin level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - C reactive protein (CRP) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the CRP level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazol
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - Creatine kinase (CK) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the CK level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - Creatinine | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the creatinine level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - Glucose (fasting) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the fasting glucose level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry- Uric acid | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the uric acid level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry- BUN | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the BUN level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - Total Bilirubin (TBL) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the TBL level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - Indirect bilirubin | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the indirect bilirubin as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - High-sensitivity troponin I ((hsTnI) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the High-sensitivity troponin I ((hsTnI) as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Serum Clinical chemistry - N-terminal-pro-brain natriuretic peptide (NT-pro-BNP) | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the N-terminal-pro-brain natriuretic peptide (NT-pro-BNP) as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.
Number of participants with abnormal laboratory assessments: Clinical Urinalysis - Protein | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the urine protein level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole. If urinalysis is positive for protein, a microscopy test will be performed to assess RBC, WBC, casts [cellular, granular, hyaline]).
Number of participants with abnormal laboratory assessments: Clinical Urinalysis - Blood | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the urine blood level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole. If urinalysis is positive for blood, a microscopy test will be performed to assess RBC, WBC, casts [cellular, granular, hyaline]).
Number of participants with abnormal laboratory assessments: Clinical Urinalysis - Glucose | From screening (Day -28) till follow-up visit (up to approximately 6 weeks)
  To assess the urine glucose level as variables of safety and tolerability after administration of single dose of AZD9977 in combination with itraconazole.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, Principal Investigator — Dr.
Locations (1):
- Research Site, Baltimore, Maryland, United States